CLINICAL TRIAL: NCT00643435
Title: Self-Efficacy Enhancing Interviewing Techniques Study
Acronym: SEE-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Anthony Jerant, MD, Department of Family and Community Medicine, UC Davis School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 200715598-1
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes; Depression; Anxiety; Asthma; Post-Traumatic Stress Disorder
Keywords: self-efficacy; chronic illness; health behavior; education, medical, residency
MeSH Terms: conditions — Diabetes Mellitus; Depression; Anxiety Disorders; Asthma; Stress Disorders, Post-Traumatic; Chronic Disease; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): These residents receive training provided by standardized patient instructors, in use of self-efficacy enhancing interviewing techniques to support patient health behavior change,
  Interventions: Behavioral: Self-efficacy enhancing interviewing techniques training
- 2 (Active Comparator): These residents receive training provided by a standardized patient instructor, regarding the common co-occurrence of chronic medical and mental health problems, without any interviewing technique discussion or training.
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: Self-efficacy enhancing interviewing techniques training — Teaching by standardized patient instructors regarding use of self-efficacy enhancing interviewing techniques to be applied in patient encounters
  Arms: 1
Behavioral: Control intervention — These residents receive training provided by a standardized patient instructor, regarding the common co-occurrence of chronic medical and mental health problems, without any interviewing technique discussion or training.
  Arms: 2

SUMMARY:
Patient self-efficacy, or confidence in one's ability to take the necessary steps to achieve a goal, has been shown to influence a number of important health behaviors and outcomes. However, current ways of increasing patient self-efficacy are time and labor intensive and occur away from doctor visits, where most health care is delivered. We developed, and are testing in a study the effectiveness of a new way of teaching doctors how to talk to patients during office visits in a way that will boost their patients' self-efficacy for changing important health behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Family medicine or internal medicine residents in training at the University of California Davis Medical Center

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Resident physician use of self-efficacy enhancing patient interviewing techniques, assessment via coding of audio recordings from standardized patient encounters | Within 6 months of completion of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anthony F Jerant, MD, Principal Investigator — Department of Family and Community Medicine, University of California Davis School of Medicine